CLINICAL TRIAL: NCT00544947
Title: Observation of Respiration Following Regional Anaesthesia With Intrathecal Opioids: a Comparison Between Diamorphine and Fentanyl Combined With Postoperative Morphine PCA Using a Carbon Dioxide Tension and Pulse Oximetry Sensor (TOSCA)
Brief Title: Observation of Respiration Following Regional Anaesthesia With Intrathecal Opioids for Caesarean Section
Status: Completed | Type: Observational
Sponsor: NHS Greater Clyde and Glasgow (Other)
Responsible Party: Dr Stephan Dalchow, NHS Greater Clyde&Glasgow
Other Study IDs: 07/S0704/67
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2009-02-04 (Estimated); Status verified 2009-02

CONDITIONS: Respiratory Depression
Keywords: Respiratory Depression; Caesarean Section; Diamorphine; Fentanyl
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- D, F: Group D will be patients at Princess Royal Maternity Hospital in Glasgow, where supplementation with intrathecal diamorphine 300mcg is the current anaesthetic technique of choice.
  Group F will be patients at the Queen Mother's Maternity Hospital in Glasgow, where supplementation with intrathecal fentanyl 15mcg plus post-operative morphine PCA is the current anaesthetic technique of choice for elective caesarean section.

SUMMARY:
Spinal Administration of opioids offers segmental analgesia, but has side effects including pruritus, nausea and vomiting, urinary retention, hypotension, and respiratory depression, both early and delayed. Many Centres in the UK now routinely use supplementation of spinal anaesthesia from bupivacaine with intrathecal fentanyl or diamorphine. If Fentanyl is used, this is usually accompanied by connection to a i.v. Morphine patient-controlled analgesia (PCA)-device in the postoperative period, whereas the use of intrathecal diamorphine seems to result in a reduction in post-operative morphine requirements, which has obviated the need for PCA devices in many centres. There has been recent controversy over which opioid is safer to use with regards to the risk of respiratory depression.1,2 The investigators want to investigate, whether intrathecal diamorphine causes less or more post-operative respiratory depression in healthy mothers undergoing elective caesarean section than intrathecal fentanyl plus post-operative morphine PCA.

DETAILED DESCRIPTION:
Method:

We will use transcutaneous carbon dioxide tension as our primary outcome measure of respiratory depression. Secondary outcome measures will be the oxygen-saturation, the respiratory rare, neurological status assessed by Glasgow Coma Scale (GCS) and the need for administration of naloxone and/or active airway management.

PtCO2 and SpO2 will be measured transcutaneously using the Linde TOSCA 500 Monitoring System, which is a relatively new miniaturized single sensor, that is applied to the earlobe.

There will be 2 study groups.

Group D will be patients at Princess Royal Maternity Hospital in Glasgow, where supplementation with intrathecal diamorphine 300mcg is the current anaesthetic technique of choice.

Group F will be patients at the Queen Mother's Maternity Hospital in Glasgow, where supplementation with intrathecal fentanyl 15mcg plus post-operative morphine PCA is the current anaesthetic technique of choice for elective caesarean section.

Additional postoperative Analgesia will be given as per local guidelines.

We will recruit 40 patients to each group.

Patients will receive verbal and written information prior to written consent before being included.

Information Gathering:

The TOSCA monitor will be connected in recovery following the end of caesarean section (with PCA connection at QMMH). Monitoring will be continuous until 0800hrs the following morning giving approx. 20 hours data for each patient.

Data will then be downloaded to a database for subsequent analysis. We will also note the total dose of morphine used in each patient and any complications that occurred or interventions carried out.

We plan to recruit an SHO on each site to help with information gathering.

Ethics Approval:

Ethics Approval has been obtained by application to the Research Ethics Committee of the Glasgow Royal Infirmary.

Statistical Analysis

For both CO2 and O2 parameters the mean area under the curve (AUC) will be compared between the diamorphine and fentanyl groups using a normal linear model. This will enable the analysis to adjust for any demographic and clinical variables, which are known to influence either of these indicators of respiratory depression.

There is no previous information in the literature on the variability in area under the curve for either CO2 concentration or O2 saturation. Any specification of effect size must therefore be in terms of a number of standard deviations, where the standard deviation is not known.

We assume that the primary endpoint is the measurement of CO2 over a period of 24 hours and that this will be quantified in the analysis using area under the curve (AUC). If we compare the mean AUC between the diamorphine and fentanyl groups using a two sample t-test (with two-sided significance level 5%) then a study including 40 patients per group would have 80% power to detect a mean AUC difference between groups of 0.634 standard deviations and 90% power to detect a mean AUC difference of and 0.851 standard deviations.

Final Statistical Analysis will be carried out in cooperation with Dr Chris Weir from the Robertson Centre for Biostatistics at the University of Glasgow.

ELIGIBILITY:
Inclusion Criteria:

* 1st patient on list
* ASA I or II
* BMI <40 at booking
* Term pregnancy +/- 2 weeks gestation

Exclusion Criteria:

* ASA>II
* BMI>40 at booking
* History of Obstructive Sleep Apnoea (OSA)
* Need for supplementation with intravenous Opioids intraoperatively
* Conversion to GA

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Elective caesarean section Healthy pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
transcutaneous carbon dioxide tension | within the first 24 hours after surgery

SECONDARY OUTCOMES:
oxygen-saturation, respiratory rate, neurological status, need for administration of naloxone and/or active airway management | within first 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Dalchow, FRCA, Principal Investigator — National Health Service
Locations (1):
- Princess Royal Maternity Hospital, Glasgow, United Kingdom